CLINICAL TRIAL: NCT02759601
Title: A Phase I/II Dose Escalation Trial of HDAC Inhibitor Tefinostat for Cancer Associated Inflamation in Hepatocellular Carcinoma
Brief Title: Dose Escalation Trial of Tefinostat for Cancer Associated Inflamation in Hepatocellular Carcinoma (HCC)
Acronym: CHR-2845
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008260QM; 2012-000326-22 (EudraCT Number)
Record Dates: First submitted 2014-10-23; First posted 2016-05-03 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: HDAC Inhibitor; Tefinostat; Inflammation; Hepatocellular Carcinoma; Cancer associated Inflammation in Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Inflammation | interventions — CHR 2845

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tefinostat (Other): This is an open label, dose escalating, phase I/II study of Tefinostat administered orally, once or twice daily in 28 day cycles of treatment in patients with advanced hepatocellular carcinoma.
  Up to 5 cohorts of 3-6 patients (number is dependent on DLT occurrence) will be treated for 28 days once or twice daily (360, 480mg once daily, then 240, 360, 480mg twice daily) to determine safety and tolerability of Tefinostat and to identify the recommended dose for Phase II.
  Interventions: Drug: Tefinostat

INTERVENTIONS:
Drug: Tefinostat — Tefinostat is a novel type of HDACi used in cancer targeted specifically to cell of monocyte - macrophase lineage

SUMMARY:
This study is being carried out to assess the best dose of a new drug, called tefinostat, in treating liver cancer.

Tefinostat is a new drug that blocks enzymes called histone deacetylases (pronounced dee-as-et-isle-azes). Cells need these enzymes to grow and divide. Blocking them may stop cancer growing. Drugs that block these enzymes are called histone deacetylase inhibitors or 'HDAC inhibitors'.

Tefinostat has never been given to patients with liver cancer before so it isn't known which dose is best at treating liver cancer. To find this out the study will be testing one dose and if that is safe, then test a higher dose and so on.

The aim of this study is to find the best dose of tefinostat without causing side effects. The study will be looking closely at any side effects patients might experience from this treatment.

DETAILED DESCRIPTION:
This is an open label, dose escalating, phase I/II study of Tefinostat administered orally, once or twice daily in 28 day cycles of treatment in patients with advanced hepatocellular carcinoma.

The starting dose of the Phase I dose escalation stage of the study has been based on the results of a previous Phase I trial of Tefinostat in patients with haematological malignancies. The starting dose of Tefinostat will be 360mg OD. As Tefinostat has a median plasma half-life of 0.47h (range 0.19 to 1.18) and CHR-2847 a median half-life of 1.4 h (range 0.98 to 3.79) twice daily dosing will also be investigated, starting at 240mg BID.

Phase I Up to 5 cohorts of 3-6 patients will be treated for 28 days once or twice daily (360, 480mg once daily, then 240, 360, 480mg twice daily) to determine safety and tolerability of Tefinostat and to identify the recommended dose for Phase II (RP2D). Patients with stable disease or with a tumour response will be allowed to continue treatment until PD or unacceptable toxicity, at the discretion of the Investigator.

Patients with advanced HCC who have not received prior systemic therapy will be eligible for the study if they are Child-Pugh classification A and are not candidates for surgical treatment, with adequate bone marrow, hepatic and renal function. Patients should not have a history of organ allograft or any serious concurrent illness.

Doses will be increased in a stepwise fashion and the decision to do so will be made by the participating Investigators on the basis of DLT, PK and PD. The starting dose will be 360mg od. Should this dose not be safe the dose level may be reduced to 240mg od. Dosing will initially take place once a day, for 28 days, while later cohorts will investigate twice daily dosing. More than one DLT in a once daily dose cohort will not preclude investigation of twice daily dosing at a lower dose.

Decisions to escalate to the next dose level, will be made jointly by the participating Investigators based on review of all the available data from the first cycle of treatment for each patient of that cohort. The first subject must have completed 7 days of the course of treatment before the next two subjects are enrolled. All subjects treated in that cohort must have undergone repeated safety evaluations prior to enrolment of the next dose cohort.

If a subject withdraws or is withdrawn from the study prior to completion of the first treatment period, in the absence of a DLT, that subject must be replaced and the replacement patient dosed at the scheduled dose, not completed, before dose escalation can occur.

Upon completion of the first treatment period of 28 days (dose finding, Phase I), suitable patients may continue with further treatment as described under Duration of Treatment, at the discretion of the investigator.

The available clinical and safety information from this trial as well as the previous single agent study of Tefinostat will be reviewed by the participating investigators, who will agree the RP2D.

The Phase I data will be reviewed by the participating investigators prior to progressing to Phase II.

Patients will be treated at the recommended phase II dose (RP2D) selected in Phase I, over an 84 day course of treatment. Approximately 39 patients with advanced HCC will be treated. Patients who have stable disease or with a tumour response after the 84 day treatment period will be allowed to continue treatment until PD or unacceptable toxicity, at the discretion of the treating investigator. Patient recruitment will continue until approximately 40 patients treated at the RP2D, including those already treated at that dose in Phase 1, are evaluable for response following treatment with at least 84 days of study therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent.
2. Histologically or cytologically confirmed malignant HCC refractory to standard therapy or for which no standard therapy exists.

   a. Patients with alcoholic cirrhosis may be included dependent on clinical judgement as to their ability to conform to the protocol.
3. Patient is not a transplant candidate.
4. Hepatitis is controlled by antiviral therapy (PEG-IFN, ribavirin, telaprevir, etc). Prophylactic Lamivudine for HBV carriers.
5. Child-Pugh classification A or B7.
6. Adequate bone marrow, hepatic and renal function including the following:

   * Hb ≥ 9.0g/dL, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥75 x 109/L.
   * Total bilirubin ≤ 1.5 x upper normal limit, excluding cases where elevated bilirubin can be attributed to Gilberts Syndrome.
   * AST (SGOT), ALT (SGPT) ≤ baseline + 4 x upper normal limit .
   * Creatinine ≤ 1.5 x upper normal limit.
   * Serum albumin > 28g/L.
   * INR < 1.5 or a Pt/PTT within normal limits.
7. Age ≥ 18 years.
8. Performance status (PS) 0-2 (ECOG scale).
9. Estimated life expectancy greater than 3 months.
10. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to start of trial. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment. Acceptable methods of contraception include IUD, oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive pessary).

Exclusion Criteria:

1. Anti-cancer therapy including chemotherapy, radiotherapy, TACE, endocrine therapy, immunotherapy or use of other investigational agents within the 4 weeks prior to trial.
2. Use of medicines known to prolong QTc within 14 days prior to the first dose of study drug (see Appendix III).
3. Candidate for surgical resection, orthotopic liver transplantation, or loco-regional therapy such as radio-frequency ablation or chemoembolization.
4. History of organ allograft.
5. Co-existing active infection or serious concurrent illness.
6. Significant cardiovascular disease as defined by:

   * History of congestive heart failure requiring therapy.
   * History of unstable angina pectoris or myocardial infarction up to 6 months prior to trial entry.
   * Presence of severe valvular heart disease.
   * Presence of a ventricular arrhythmia requiring treatment.
   * LVEF < 50% (or less than institutional norm- some places have 45%).
   * QTc interval ≥ 450ms for men and ≥ 470ms for women (using Bazett's formula).
7. Any co-existing medical condition that in the Investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
8. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies.
9. Gastrointestinal disorders that may interfere with absorption of the study drug.
10. Patients requiring palliative radiotherapy within the last 4 weeks of study entry.
11. Uncontrolled hypercalcaemia (>CTCAE v4.03 grade I).
12. Pregnant or breast-feeding women.
13. Patients who have received an investigational drug within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose | For 28 days following commencing IMP treatment. (Phase I)
  Determining the maximal dose at either once or twice daily dosing at which no more than one patient (out of 3) at that dose level experiences a DLT.

SECONDARY OUTCOMES:
Response Assessment | From registration to disease progression.
  Response assessment (stable disease (SD), partial response (PR) or complete response (CR)) determined according to modified Response Evaluation Criteria in Solid Tumours (mRECIST v1.1) in all patients receiving at least one cycle of treatment. Response assessment should take place at 1 month and then again after every 2 months of further treatment.
Phase I & II: To determine pharmacokinetic parameters for tefinostat and CHR-2847 when administered orally at different dose levels and dose schedules. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  Measurement of PK parameter values for tefinostat and CHR-2847 on day 1 and day 28 of the 1st cycle, using PK profiles generated from samples taken at the protocol specified time points.

OTHER OUTCOMES:
Phase I & II: To assess responses to target inhibition by tefinostat. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  Inhibition of target genes and microarray target gene responses in tumour biopsies and peripheral blood monocytes.
Phase I & II: The impact of HDACi on circulating cytokine profiles. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  Ex vivo analysis of plasma using the Meso Scale Discovery (MSD) platform, correlation to disease status and response.
Phase I & II: To explore the feasibility of measuring tefinostat levels in tumour tissue. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  Measurement of tissue concentrations of tefinostat.
Phase I & II: To establish relationships between measures of tumour expression of hCE-1 and objective tumour response. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  hCE-1 expression in liver biopsies will be quantified by IHC. Correlation between presence/absence of hCE-1 versus objective tumour response will be analysed.
Phase I & II: To explore Enhanced Liver Function (ELF) test to monitor liver toxicity under tefinostat. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  The combination of HA, P3NP and TIMP-1 measured by ELISA be used to determine the severity of liver fibrosis with good accuracy (Rosenberg et al, 2004).
Phase I & II: To determine the impact of HDACi on anti-tumour immune responses. | Phase I: End of 28 day treatment period; Phase II: End of 84 days period
  Serial assessment of TAA-specific CTLs in peripheral blood using EliSPOT, gamma capture and multimer assays (and, where feasible, on T cells from serial tumour biopsies).

CONTACTS AND LOCATIONS:
Overall Officials: David Propper, Principal Investigator — Barts NHS Trust
Locations (4):
- United Kingdom (4):
  - Barts Health NHS Trust, London, Greater London
  - Beatson Cancer Centre, Glasgow
  - Clatterbridge Cancer Centre, Liverpool
  - University College London Hospital, London